CLINICAL TRIAL: NCT06711042
Title: The Effect of Spinopelvic Movements on Hip Functions in Patients With Total Hip Arthroplasty
Brief Title: How Spinopelvic Movements Affect Hip Function After Total Hip Arthroplasty
Acronym: THA
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Elif AYGUN POLAT, PhD, Ordu University
Other Study IDs: ODU-SBFTR-AYGUNPOLAT-004
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Total Hip Replacement; Hip Dislocation; Hip Osteoarthritis
MeSH Terms: conditions — Hip Dislocation; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group (Implant Placement Within Functional Safe Zone - FSZ): This group will consist of patients who have previously undergone total hip arthroplasty (TKA) with implant placement within the functional safe zone (FSZ).
  Interventions: Diagnostic Test: functional tests and radiographic analysis
- Experimental Group (Implant Placement Outside Functional Safe Zone - FSZ): This group will consist of patients who have previously undergone total hip arthroplasty (TKA) but have implant placement outside the functional safe zone (FSZ).
  Interventions: Diagnostic Test: functional tests and radiographic analysis

INTERVENTIONS:
Diagnostic Test: functional tests and radiographic analysis — In this observational study, no active interventions or treatments will be administered to the participants. Both groups (Control Group and Experimental Group) will undergo clinical evaluations, including functional tests (WOMAC, Harris Hip Score, Oxford Hip Score, SF-12, TUG) and radiographic analysis (angular measurements). The participants' outcomes will be compared based on their implant placement (within or outside the Functional Safe Zone).

SUMMARY:
Our study aims to evaluate the effect of spinopelvic movement on hip functions in individuals who have undergone total hip arthroplasty (THA). This study will contribute to the literature by helping identify and prevent issues experienced by THA patients, ranging from hip pain to limited mobility and even hip dislocation.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a widely accepted surgical procedure that effectively alleviates pain, enhances mobility, and improves physical function in patients with hip osteoarthritis. However, improper placement of implants during surgery can lead to complications such as abnormal edge loading, early wear of polyethylene components, ceramic insert fractures, or hip dislocations, often requiring early revision surgeries. While Lewinnek's "safe zone" (30°-50° inclination and 5°-25° anteversion for the acetabular component) has traditionally been used as a guideline, recent studies have reported significant dislocation rates even within these parameters, highlighting spinopelvic movement abnormalities as a critical factor. Normal spinopelvic-hip mechanics allow for adaptive changes in the pelvis and acetabulum during positional transitions, thereby preventing anterior or posterior impingement in the hip joint. However, patients with restricted lumbosacral mobility are at a greater risk of impingement-related symptoms. To address these challenges, advanced metrics such as sacral slope difference (ΔSS), pelvic-femoral angle (PFA), and combined sagittal index (CSI) have been introduced to better define functional safe zones and assess risks of hip impingement and dislocation. While the relationship between CSI and hip dislocations is established, its impact on hip function remains unclear. This study aims to evaluate the effect of spinopelvic movement on hip function in individuals who have undergone THA. By identifying and preventing complications such as hip pain, mobility restrictions, and dislocations, the research seeks to provide meaningful contributions to the literature and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 and older.
* At least 12 months post-surgery.

Exclusion Criteria:

* Patients with modular neck implants, metal-metal, or ceramic bearing surfaces.
* Patients with hip infection or advanced osteoarthritis in the contralateral hip.
* Patients with leg length discrepancy.
* Patients with neurological, orthopedic, or systemic diseases affecting gait or balance.
* Patients with a body mass index (BMI) greater than 40 kg/m².

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients who underwent primary total hip arthroplasty using the posterolateral approach by the same surgeon at Ordu University Training and Research Hospital, Department of Orthopedics and Traumatology, during the years 2022-2023. Eligible patients must be aged 60 years or older and have a minimum of 12 months post-surgery.
  Exclusion criteria include patients with modular neck implants, metal-metal, or ceramic bearing surfaces, hip infections, advanced osteoarthritis in the contralateral hip, leg length discrepancy, neurological, orthopedic, or systemic diseases affecting gait or balance, or a body mass index (BMI) greater than 40 kg/m².
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Radiographic Angular Measurements | At least 12 months after surgery
  The angular measurements of the implant positions will be assessed using pre-existing routine control radiographs. This includes analysis of the pelvic tilt, acetabular anteversion, and femoral anteversion, which will be measured by two experienced radiologists using the General Electric Centricity PACS system.
WOMAC (Western Ontario and McMaster Osteoarthritis Index) | At least 12 months after surgery
  The WOMAC score will be used to assess pain, stiffness, and physical function in patients with hip osteoarthritis. It includes 24 questions across three domains: pain, stiffness, and physical function
Harris Hip Score (HHS) | At least 12 months after surgery
  The Harris Hip Score will be used to assess the hip function and pain level in patients who have undergone total hip arthroplasty. It consists of several domains, including pain, function, range of motion, and deformity.
Oxford Hip Score | At least 12 months after surgery
  The Oxford Hip Score will be used to assess hip function and the impact of hip arthritis on patients' quality of life. It includes questions on pain and function during daily activities.
SF-12 (Short Form-12 Health Survey) | At least 12 months after surgery
  The SF-12 is a 12-item questionnaire used to assess the overall health-related quality of life. It includes physical and mental health components and provides a summary score for each.
TUG (Timed Up and Go) Test | At least 12 months after surgery
  The Timed Up and Go (TUG) test is a functional assessment to evaluate mobility, balance, and risk of falls. The patient is asked to rise from a seated position, walk 3 meters, turn around, walk back, and sit down again. The total time taken to complete the task is measured in seconds. It is useful in assessing recovery progress and mobility after total hip arthroplasty (THA).

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf POLAT, Assoc.Prof., Study Director — Ordu University; Elif AYGUN POLAT, PhD, Principal Investigator — Ordu University; Murat ALPARSLAN, MD, Principal Investigator — Ordu University; Tolga KECECİ, Assoc.Prof., Principal Investigator — Ordu University; Alper ÇIRAKLI, Prof., Study Chair — Ordu University
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No